CLINICAL TRIAL: NCT01645475
Title: Desmopressin Melt: Impact on Sleep and Daytime Functioning? A Prospective Study.
Brief Title: Desmopressin Melt: Impact on Sleep and Daytime Functioning
Acronym: SLEEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/247
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2014-12

CONDITIONS: Monosymptomatic Nocturnal Enuresis
Keywords: enuresis
MeSH Terms: conditions — Enuresis | interventions — Freezing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin lyophilisate (Melt) (Experimental): Patients receiving Desmopressin lyophilisate (Melt).
  Interventions: Drug: Desmopressin lyophilisate (Melt)

INTERVENTIONS:
Drug: Desmopressin lyophilisate (Melt) — Patient receives Desmopressin lyophilisate (Melt).

SUMMARY:
Nocturnal enuresis affects 10% of the 7-year-old children and is essentially caused by a mismatch between nocturnal bladder capacity and the amount of urine produced during the night together with failure of the child to awaken in response to a full bladder.Urine overproduction at night or nocturnal polyuria (NP) is a major factor contributing to monosymptomatic nocturnal enuresis (MNE) pathophysiology in a large proportion of patients.

Since NP is related to an abnormal circadian rhythm of arginine vasopressin (AVP) secretion, the synthetic AVP analogue desmopressin is widely used to treat MNE.

It is recommended by the International Consultation on Incontinence (grade A,level 1). Desmopressin is available in 3 different formulations: nasal spray, tablet and the newest form melt.

Baeyens et al demonstrated an increased prevalence of attention deficit-hyperactivity disorder (ADHD) in children with MNE According to recent data there is a high incidence of periodic limb movements in sleep at night in children with nocturnal enuresis. Those children have an increased cortical arousability leading to awakening.

The frequent awakening most likely has an influence on concentration and other ADHD-symptoms in daily life.

This study will assess the impact of desmopressin melt on prepulse inhibition, ADHD-symptoms, cognition and learning, sleep, quality of life and self esteem.

New patients aged 6-16 years with monosymptomatic nocturnal enuresis, nocturnal polyuria and sleep problems are tested before the start of the study medication desmopressin melt (T1) and 6 months later (T2). It is a multi-method, multi-informant study.

ELIGIBILITY:
Inclusion Criteria:

* New patient
* age 6 to 16 years
* monosymptomatic nocturnal enuresis, nocturnal polyuria and sleep problems

Exclusion Criteria:

* mental retardation
* autism spectrum disorders
* daytime incontinence resistant to therapy
* dysfunctional voiding
* poor therapy-compliance
* diuretics, antihypertensives, uropathy, renal abnormalities

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bladder information: voiding calender | Change between day 1 before start of studymedication and 6 months later
  Voiding calendar
Urine concentration | Change between day 1 before start of studymedication and 6 months later
  Forced diuresis and 24h concentration profile with measurement of Na, K, creatinin, osmolality
IQ (Intelligent Quotient) | Change between day 1 before start of studymedication and 6 months later
  Wechsler Intelligence Scale for Children-Third Edition (WISC-III) short version
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Child Behavior Checklist - CBCL (parents)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  "Vragenlijst voor Gedragsproblemen bij Kinderen" (VvGK): questionnaire to screen for ADHD and behavioral disorders (parents, teacher)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  TRF: Teacher Report Form (teacher)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Behavior Rating Inventory of Executive Function (BRIEF): questionnaire to assess executive functions) (parents, teacher)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Pediatric Incontinence Questionniare (PinQ): questionnaire to measure health related quality of life, specific enuresis (parents + child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Pediatric Quality of Life Inventory (PedsQL): questionnaire to measure health related quality of life (parents + child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Kiddie Schedule for Affective Disorders and Schizofrenia (K-SADS): diagnostic interview if CBCL/TRF is (sub)clinical (parents + child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Cambridge Neuropsychological Test Automated Battery (CANTAB) (child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  IQ: WISC-III subtest Digit Span - children are orally given sequences of numbers and asked to repeat them, either as heard or in reverse order. (child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Test of Everyday Attention for Children (TEA-ch): subtest Secret code + Score DT (sustained attention task) (child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  "Competentiebelevingsschaal voor Kinderen/Adolescenten" (CBSK/CBSA): questionnaire to measure self-esteem in children or adolescents OR The pictorial scale of perceived competence and social acceptance for young children. (child)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  Swanson, Kotkin, Agler, Mylnn, and Pelham (SKAMP) Rating Scale: observation scale (teacher)
Psychological functioning questionnaire | Change between day 1 before start of studymedication and 6 months later
  School results: copy of schoolreport (+median) (teacher)
Sleep | Change between day 1 before start of studymedication and 6 months later
  Pediatric Sleep Questionnaire (questionnaire to assess the quality of sleep) (parents)
Sleep | Change between day 1 before start of studymedication and 6 months later
  Children's Sleep Habits Questionnaire (CSHQ) (parents)
Sleep | Change between day 1 before start of studymedication and 6 months later
  Polysomnography (overnight hospitalization) (child)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vande Walle, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Van Herzeele C, Dhondt K, Roels SP, Raes A, Hoebeke P, Groen LA, Vande Walle J. Desmopressin (melt) therapy in children with monosymptomatic nocturnal enuresis and nocturnal polyuria results in improved neuropsychological functioning and sleep. Pediatr Nephrol. 2016 Sep;31(9):1477-84. doi: 10.1007/s00467-016-3351-3. Epub 2016 Apr 11. PMID 27067081
- See also: Related Info — http://www.uzgent.be